CLINICAL TRIAL: NCT03517618
Title: A Phase II Study Assessing Efficacy and Safety of TS-1 in Combination With Calcium Folinate in Patients With Heavily Pre-treated Metastatic Colorectal Cancer
Brief Title: TS-1 in Combination With Calcium Folinate in Patients With Heavily Pre-treated mCRC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: TTY Biopharm (Industry)
Collaborators: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TG1307
Record Dates: First submitted 2018-04-12; First posted 2018-05-07 (Actual); Last update posted 2018-05-07 (Actual); Status verified 2018-04

CONDITIONS: Metastatic Colorectal Cancer
Keywords: A phase II study; Heavily pre-treated metastatic colorectal cancer; S-1; oral leucovrin
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- S-1 + leucovorin (Experimental): Single arm
  Interventions: Drug: S-1+leucovorin

INTERVENTIONS:
Drug: S-1+leucovorin — Eligible patients will receive TS-1 orally 40-60 mg (depending on patient's body surface area (BSA)) in combination with calcium folinate 30 mg twice a day for 7 days in a 2-week cycle.
  The treatment will be administered until disease progression, intolerable toxicity, or consent withdrawal during any time of the study.
  Other Names: TS-1+calcium folinate

SUMMARY:
Primary Objective:

To determine disease control rate (DCR) of TS-1® in patients with heavily pre-treated metastatic colorectal cancer

Secondary Objectives:

* To determine objective response rate (ORR)
* To determine time to progression (TTP)
* To determine overall survival (OS)
* To assess incidence of adverse events (AEs), serious adverse events (SAEs) [Safety and Tolerability]

DETAILED DESCRIPTION:
Simon's optimal two-stage design will be used to determine the sample size for this study.

• Stage I: >1/9: The first 9 evaluable patients enrolled, >1 (or ≥2) responders are required in order to enter the second stage, otherwise the trial will be terminated at the first stage due to futility.

• Stage II: Total >8/34: For the total 34 evaluable patients, >8 (or ≥9) responders are required to conclude the effectiveness of the study regimen.

The primary endpoint will be disease control rate which will be presented in frequency tabulation with two-sided 95% confidence interval (using binomial estimation).

The secondary endpoints are described as follows:

* ORR will be presented in frequency tabulation with two-sided 95% confidence interval;
* TTP will be estimated by Kaplan-Meier method with two-sided 95% confidence interval;
* OS will be estimated by Kaplan-Meier method with two-sided 95% confidence interval;
* Incidence of adverse events (AEs), serious adverse events (SAEs) [Safety and Tolerability] : assessed by CTCAE v4.0. Safety parameters will only be analyzed on the safety analysis set and be presented in frequency tabulation.

ELIGIBILITY:
Inclusion Criteria:

1. histologically or cytologically confirmed colorectal adenocarcinoma;
2. metastatic and unresectable disease;
3. presence of at least one measurable tumor lesion which is defined as lesion that can be measured in at least one dimension (longest diameter) with a minimum size of:

   1. 10mm by CT scan and MRI (no less than double the slice thickness and a minimum of 10mm);
   2. 20mm by conventional techniques;
4. previously treatment to

   1. fluoropyrimidine, oxaliplatin and irinotecan;
   2. at least one targeted therapy
5. adequate hematopoietic function which is defined as below:

   1. hemoglobin ≥ 9 g/dL;
   2. absolute neutrophil count (ANC) ≥ 1,500/mm3;
   3. platelet count ≥ 100,000/mm3;
6. adequate hepatic function which is defined as below:

   1. total bilirubin ≤ 2 times upper limit of normal (ULN);
   2. hepatic transaminases (ALT and AST) ≤ 3 x ULN. If there are known liver metastases, ALT or AST must be ≤ 5 x ULN;
7. adequate renal function which is defined as below:

   a. serum creatinine ≤ 1.5 x ULN;
8. age of 20 years or above;
9. ECOG performance status 0-2;
10. life expectancy of at least 12 weeks;
11. ability to take oral medication;
12. ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria:

1. history or known presence of brain metastasis;
2. presence of mental disease or psychotic manifestation;
3. significant medical conditions that is contraindicated to study medication or render patient at high risk from treatment complications based on investigator's discretion;
4. presence of diarrhea ≥ grade 2 in common terminology criteria for adverse event version 4.0 (CTCAE v4.0);
5. other malignancy within the past 5 years (different site or histology) except for adequately treated basal or squamous cell skin cancer or cervical cancer in situ;
6. recent (within 30 days prior to study treatment) treatment of another investigational drug;
7. pregnant women or nursing mothers, or positive pregnancy test for women of childbearing potential. Patients with childbearing potential should have effective contraception for both the patient and his or her partner during the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2014-07-05 (Actual); Primary Completion 2015-06-18 (Actual); Study Completion 2015-06-18 (Actual)

PRIMARY OUTCOMES:
Disease Control Rate (DCR) | 6 months(an expected average)
  Documented objective response (OR) (defined as partial response [PR] or complete response [CR]), assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 at any time during trial participation by Investigator assessment

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 6 months(an expected average)
  the rate of completely response [CR] and partial response [PR] patients according to RECIST version 1.1. criteria
Time to Progression (TTP) | until disease progression, intolerable toxicity, 12 months(an expected average)
  Participants follow-up for disease progression occur. Maximum follow-up time is 12 months after the initial administration of the last subject
Overall survival (OS) | at death or at the end of study, 24 months(an expected average)
  median time between the start date of study treatment and the date of the death
Incidence of adverse events (AEs), serious adverse events (SAEs) [Safety and Tolerability] | From the date of study entry until 30 days after the last dose of study treatment
  assessed by the NCI-CTCAE (Common Toxicity Criteria for Adverse Effects) v4.0 and within some subgroups of patients

CONTACTS AND LOCATIONS:
Overall Officials: Hung-Chih Hsu, Principal Investigator — Chang Gung Memorial Hospital, Linkou, Taiwan
Locations (1):
- Chang-Gung Memorial Hospital, Linkou, Linkou District, Taiwan

REFERENCES:
- [Background] Lee WS, Yun SH, Chun HK, Lee WY, Yun HR, Kim J, Kim K, Shim YM. Pulmonary resection for metastases from colorectal cancer: prognostic factors and survival. Int J Colorectal Dis. 2007 Jun;22(6):699-704. doi: 10.1007/s00384-006-0218-2. Epub 2006 Nov 16. PMID 17109105
- [Background] Van Cutsem E, Nordlinger B, Adam R, Kohne CH, Pozzo C, Poston G, Ychou M, Rougier P; European Colorectal Metastases Treatment Group. Towards a pan-European consensus on the treatment of patients with colorectal liver metastases. Eur J Cancer. 2006 Sep;42(14):2212-21. doi: 10.1016/j.ejca.2006.04.012. Epub 2006 Aug 10. PMID 16904315
- [Background] Yoo PS, Lopez-Soler RI, Longo WE, Cha CH. Liver resection for metastatic colorectal cancer in the age of neoadjuvant chemotherapy and bevacizumab. Clin Colorectal Cancer. 2006 Sep;6(3):202-7. doi: 10.3816/CCC.2006.n.036. PMID 17026789
- [Background] Alberts SR, Horvath WL, Sternfeld WC, Goldberg RM, Mahoney MR, Dakhil SR, Levitt R, Rowland K, Nair S, Sargent DJ, Donohue JH. Oxaliplatin, fluorouracil, and leucovorin for patients with unresectable liver-only metastases from colorectal cancer: a North Central Cancer Treatment Group phase II study. J Clin Oncol. 2005 Dec 20;23(36):9243-9. doi: 10.1200/JCO.2005.07.740. Epub 2005 Oct 17. PMID 16230673
- [Background] Dawood O, Mahadevan A, Goodman KA. Stereotactic body radiation therapy for liver metastases. Eur J Cancer. 2009 Nov;45(17):2947-59. doi: 10.1016/j.ejca.2009.08.011. Epub 2009 Sep 19. PMID 19773153
- [Background] Kemeny N. Management of liver metastases from colorectal cancer. Oncology (Williston Park). 2006 Sep;20(10):1161-76, 1179; discussion 1179-80, 1185-6. PMID 17024869
- [Background] Muratore A, Zorzi D, Bouzari H, Amisano M, Massucco P, Sperti E, Capussotti L. Asymptomatic colorectal cancer with un-resectable liver metastases: immediate colorectal resection or up-front systemic chemotherapy? Ann Surg Oncol. 2007 Feb;14(2):766-70. doi: 10.1245/s10434-006-9146-1. Epub 2006 Nov 14. PMID 17103261
- [Background] Andre T, Louvet C, Maindrault-Goebel F, Couteau C, Mabro M, Lotz JP, Gilles-Amar V, Krulik M, Carola E, Izrael V, de Gramont A. CPT-11 (irinotecan) addition to bimonthly, high-dose leucovorin and bolus and continuous-infusion 5-fluorouracil (FOLFIRI) for pretreated metastatic colorectal cancer. GERCOR. Eur J Cancer. 1999 Sep;35(9):1343-7. doi: 10.1016/s0959-8049(99)00150-1. PMID 10658525
- [Background] Jager E, Heike M, Bernhard H, Klein O, Bernhard G, Lautz D, Michaelis J, Meyer zum Buschenfelde KH, Knuth A. Weekly high-dose leucovorin versus low-dose leucovorin combined with fluorouracil in advanced colorectal cancer: results of a randomized multicenter trial. Study Group for Palliative Treatment of Metastatic Colorectal Cancer Study Protocol 1. J Clin Oncol. 1996 Aug;14(8):2274-9. doi: 10.1200/JCO.1996.14.8.2274. PMID 8708717
- [Background] Falcone A, Ricci S, Brunetti I, Pfanner E, Allegrini G, Barbara C, Crino L, Benedetti G, Evangelista W, Fanchini L, Cortesi E, Picone V, Vitello S, Chiara S, Granetto C, Porcile G, Fioretto L, Orlandini C, Andreuccetti M, Masi G; Gruppo Oncologico Nord Ovest. Phase III trial of infusional fluorouracil, leucovorin, oxaliplatin, and irinotecan (FOLFOXIRI) compared with infusional fluorouracil, leucovorin, and irinotecan (FOLFIRI) as first-line treatment for metastatic colorectal cancer: the Gruppo Oncologico Nord Ovest. J Clin Oncol. 2007 May 1;25(13):1670-6. doi: 10.1200/JCO.2006.09.0928. PMID 17470860
- [Background] Souglakos J, Androulakis N, Syrigos K, Polyzos A, Ziras N, Athanasiadis A, Kakolyris S, Tsousis S, Kouroussis Ch, Vamvakas L, Kalykaki A, Samonis G, Mavroudis D, Georgoulias V. FOLFOXIRI (folinic acid, 5-fluorouracil, oxaliplatin and irinotecan) vs FOLFIRI (folinic acid, 5-fluorouracil and irinotecan) as first-line treatment in metastatic colorectal cancer (MCC): a multicentre randomised phase III trial from the Hellenic Oncology Research Group (HORG). Br J Cancer. 2006 Mar 27;94(6):798-805. doi: 10.1038/sj.bjc.6603011. PMID 16508637
- [Background] Cassidy J, Clarke S, Diaz-Rubio E, Scheithauer W, Figer A, Wong R, Koski S, Lichinitser M, Yang TS, Rivera F, Couture F, Sirzen F, Saltz L. Randomized phase III study of capecitabine plus oxaliplatin compared with fluorouracil/folinic acid plus oxaliplatin as first-line therapy for metastatic colorectal cancer. J Clin Oncol. 2008 Apr 20;26(12):2006-12. doi: 10.1200/JCO.2007.14.9898. PMID 18421053
- [Background] Petrelli N, Herrera L, Rustum Y, Burke P, Creaven P, Stulc J, Emrich LJ, Mittelman A. A prospective randomized trial of 5-fluorouracil versus 5-fluorouracil and high-dose leucovorin versus 5-fluorouracil and methotrexate in previously untreated patients with advanced colorectal carcinoma. J Clin Oncol. 1987 Oct;5(10):1559-65. doi: 10.1200/JCO.1987.5.10.1559. PMID 2443619
- [Background] Wolmark N, Rockette H, Fisher B, Wickerham DL, Redmond C, Fisher ER, Jones J, Mamounas EP, Ore L, Petrelli NJ, et al. The benefit of leucovorin-modulated fluorouracil as postoperative adjuvant therapy for primary colon cancer: results from National Surgical Adjuvant Breast and Bowel Project protocol C-03. J Clin Oncol. 1993 Oct;11(10):1879-87. doi: 10.1200/JCO.1993.11.10.1879. PMID 8410113
- [Background] Cassidy J, Tabernero J, Twelves C, Brunet R, Butts C, Conroy T, Debraud F, Figer A, Grossmann J, Sawada N, Schoffski P, Sobrero A, Van Cutsem E, Diaz-Rubio E. XELOX (capecitabine plus oxaliplatin): active first-line therapy for patients with metastatic colorectal cancer. J Clin Oncol. 2004 Jun 1;22(11):2084-91. doi: 10.1200/JCO.2004.11.069. PMID 15169795
- [Background] Porschen R, Arkenau HT, Kubicka S, Greil R, Seufferlein T, Freier W, Kretzschmar A, Graeven U, Grothey A, Hinke A, Schmiegel W, Schmoll HJ; AIO Colorectal Study Group. Phase III study of capecitabine plus oxaliplatin compared with fluorouracil and leucovorin plus oxaliplatin in metastatic colorectal cancer: a final report of the AIO Colorectal Study Group. J Clin Oncol. 2007 Sep 20;25(27):4217-23. doi: 10.1200/JCO.2006.09.2684. Epub 2007 Jun 4. PMID 17548840
- [Background] Sargent DJ, Kohne CH, Sanoff HK, Bot BM, Seymour MT, de Gramont A, Porschen R, Saltz LB, Rougier P, Tournigand C, Douillard JY, Stephens RJ, Grothey A, Goldberg RM. Pooled safety and efficacy analysis examining the effect of performance status on outcomes in nine first-line treatment trials using individual data from patients with metastatic colorectal cancer. J Clin Oncol. 2009 Apr 20;27(12):1948-55. doi: 10.1200/JCO.2008.20.2879. Epub 2009 Mar 2. PMID 19255311
- [Background] Chibaudel B, Tournigand C, Andre T, de Gramont A. Therapeutic strategy in unresectable metastatic colorectal cancer. Ther Adv Med Oncol. 2012 Mar;4(2):75-89. doi: 10.1177/1758834011431592. PMID 22423266
- [Background] Lievre A, Bachet JB, Boige V, Cayre A, Le Corre D, Buc E, Ychou M, Bouche O, Landi B, Louvet C, Andre T, Bibeau F, Diebold MD, Rougier P, Ducreux M, Tomasic G, Emile JF, Penault-Llorca F, Laurent-Puig P. KRAS mutations as an independent prognostic factor in patients with advanced colorectal cancer treated with cetuximab. J Clin Oncol. 2008 Jan 20;26(3):374-9. doi: 10.1200/JCO.2007.12.5906. PMID 18202412
- [Background] Grothey A, Sargent D, Goldberg RM, Schmoll HJ. Survival of patients with advanced colorectal cancer improves with the availability of fluorouracil-leucovorin, irinotecan, and oxaliplatin in the course of treatment. J Clin Oncol. 2004 Apr 1;22(7):1209-14. doi: 10.1200/JCO.2004.11.037. PMID 15051767
- [Background] Ohtsu A, Baba H, Sakata Y, Mitachi Y, Horikoshi N, Sugimachi K, Taguchi T. Phase II study of S-1, a novel oral fluorophyrimidine derivative, in patients with metastatic colorectal carcinoma. S-1 Cooperative Colorectal Carcinoma Study Group. Br J Cancer. 2000 Jul;83(2):141-5. doi: 10.1054/bjoc.2000.1236. PMID 10901361
- [Background] Shirao K, Ohtsu A, Takada H, Mitachi Y, Hirakawa K, Horikoshi N, Okamura T, Hirata K, Saitoh S, Isomoto H, Satoh A. Phase II study of oral S-1 for treatment of metastatic colorectal carcinoma. Cancer. 2004 Jun 1;100(11):2355-61. doi: 10.1002/cncr.20277. PMID 15160338
- [Background] Van den Brande J, Schoffski P, Schellens JH, Roth AD, Duffaud F, Weigang-Kohler K, Reinke F, Wanders J, de Boer RF, Vermorken JB, Fumoleau P. EORTC Early Clinical Studies Group early phase II trial of S-1 in patients with advanced or metastatic colorectal cancer. Br J Cancer. 2003 Mar 10;88(5):648-53. doi: 10.1038/sj.bjc.6600781. PMID 12659110
- [Background] Jeung HC, Rha SY, Cho BC, Yoo NC, Roh JK, Roh WJ, Chung HC, Ahn JB. A phase II trial of S-1 monotherapy in metastatic colorectal cancer after failure of irinotecan- and oxaliplatin-containing regimens. Br J Cancer. 2006 Dec 18;95(12):1637-41. doi: 10.1038/sj.bjc.6603468. Epub 2006 Nov 14. PMID 17106441
- [Background] Lee DJ, Lee J, Lee HY, Lim T, Lee SJ, Yi SY, Park SH, Park JO, Lim HY, Kang WK, Park YS. Salvage S-1 monotherapy in metastatic colorectal cancer patients who failed irinotecan-based or oxaliplatin-based chemotherapy. Med Oncol. 2011 Dec;28 Suppl 1:S291-4. doi: 10.1007/s12032-010-9755-1. Epub 2010 Nov 30. PMID 21116875
- [Background] Yamada Y, Tahara M, Miya T, Satoh T, Shirao K, Shimada Y, Ohtsu A, Sasaki Y, Tanigawara Y. Phase I/II study of oxaliplatin with oral S-1 as first-line therapy for patients with metastatic colorectal cancer. Br J Cancer. 2008 Mar 25;98(6):1034-8. doi: 10.1038/sj.bjc.6604271. Epub 2008 Mar 4. PMID 18319719
- [Background] Kim SY, Hong YS, Kim BC, Park JW, Choi HS, Jeong SY, Kim DY, Hong CW, Sohn DK, Jung KH. A phase II study of S-1 plus irinotecan and oxaliplatin in heavily-treated patients with metastatic colorectal cancer. Invest New Drugs. 2009 Jun;27(3):269-74. doi: 10.1007/s10637-008-9177-5. Epub 2008 Sep 25. PMID 18815728
- [Background] Muro K, Boku N, Shimada Y, Tsuji A, Sameshima S, Baba H, Satoh T, Denda T, Ina K, Nishina T, Yamaguchi K, Takiuchi H, Esaki T, Tokunaga S, Kuwano H, Komatsu Y, Watanabe M, Hyodo I, Morita S, Sugihara K. Irinotecan plus S-1 (IRIS) versus fluorouracil and folinic acid plus irinotecan (FOLFIRI) as second-line chemotherapy for metastatic colorectal cancer: a randomised phase 2/3 non-inferiority study (FIRIS study). Lancet Oncol. 2010 Sep;11(9):853-60. doi: 10.1016/S1470-2045(10)70181-9. Epub 2010 Aug 12. PMID 20708966
- [Background] Hong YS, Park YS, Lim HY, Lee J, Kim TW, Kim KP, Kim SY, Baek JY, Kim JH, Lee KW, Chung IJ, Cho SH, Lee KH, Shin SJ, Kang HJ, Shin DB, Jo SJ, Lee JW. S-1 plus oxaliplatin versus capecitabine plus oxaliplatin for first-line treatment of patients with metastatic colorectal cancer: a randomised, non-inferiority phase 3 trial. Lancet Oncol. 2012 Nov;13(11):1125-32. doi: 10.1016/S1470-2045(12)70363-7. Epub 2012 Oct 10. PMID 23062232
- [Background] Koizumi W, Boku N, Yamaguchi K, Miyata Y, Sawaki A, Kato T, Toh Y, Hyodo I, Nishina T, Furuhata T, Miyashita K, Okada Y. Phase II study of S-1 plus leucovorin in patients with metastatic colorectal cancer. Ann Oncol. 2010 Apr;21(4):766-771. doi: 10.1093/annonc/mdp371. Epub 2009 Oct 14. PMID 19828562